CLINICAL TRIAL: NCT00576862
Title: Multicenter,Open,Uncontrolled,Clinical Extension Trial in Subjects With Type I Diabetes Previously Participating in Study HMR1964A/3011 in Belgium
Brief Title: Extension to Study HMR1964A/3011 in Belgium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4046
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — The subjects will continue the treatment with HOE 901 in the same way as they have done in the previous study. Based on the investigator's assessment and the approved SPC in Belgium/Luxembourg, the dosage can be adjusted individually. HOE 901 is to be injected once daily. HOE 901 must not be mixed with any other insulin, including regular human insulin or fast-acting insulin analogues.

SUMMARY:
The purpose of this trial is to allow patients to continue on HOE 901 until launch and to gather additional long-term safety data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects treated with HOE901 and who, in the judgement of the investigator, have benefited from the use of HOE 901 in a previous clinical study with HOE 901.
* Subjects treated with HOE 901 in a previous clinical study with HOE 901 for whom a change of basal insulin would destabilise glucose metabolism.
* Subjects who are likely to comply with the investigator's instructions.

Exclusion Criteria:

* Evidence of an uncooperative attitude.
* Subject not on adequate contraception, or who is pregnant, or breast feeding.
* Subject unable to understand informed consent.
* Patient receiving or likely to receive HOE901 treatment outside of SPC or PI recommendations.
* Subject becomes pregnant or is planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Evolution of efficacy parameters between first study visit (V1) and last study visit (V5) | Mean time interval: 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Elke Meyssen, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Brussels, Belgium